CLINICAL TRIAL: NCT04439084
Title: COVID-19 in Patients With Chronic Liver Diseases
Acronym: COLD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 55819
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Chronic Liver Disease
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Liver Disease Group: COVID-19 patients with Chronic Liver Disease.
  Interventions: Other: Prospective Chart Review
- Control Group: COVID-19 patients without Chronic Liver Disease.
  Interventions: Other: Prospective Chart Review

INTERVENTIONS:
Other: Prospective Chart Review — Collected data will include demographic features, clinical characteristics, clinical outcome, medication use, COVID-19-related complications in patients with chronic liver disease.

SUMMARY:
This study seeks to determine how COVID-19 affects the clinical outcome of patients with chronic liver disease, and whether the clinical course of COVID-19 is influenced by underlying chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19
* Personal history of either

  * Chronic hepatitis C
  * Chronic hepatitis B
  * Alcoholic liver disease
  * Non alcoholic liver disease
  * Autoimmune hepatitis, Primary biliary cholangitis, Primary sclerosing cholangitis
  * Cryptogenic cirrhosis
  * Hepatocellular carcinoma

Exclusion Criteria:

* Non-COVID-19 patient

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease with a confirmed diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 30 days
  Death due to any cause
All-cause mortality | 1 year
  Death due to any cause
Liver-related mortality | 28 days
  Death due to liver-related cause
Liver-related mortality | 1 year
  Death due to liver-related cause
Overall survival | Up to 1 year
  Patients will be assessed for this outcome for up to 1 year
Number of patients with hepatic decompensation | Up to 1 year
  Onset of hepatic decompensation due to COVID-19 disease; patients will be assessed for this outcome for up to 1 year

SECONDARY OUTCOMES:
Number of patients requiring hospitalization | Up to 1 year
  Patients will be assessed for this outcome for up to 1 year.
Duration of hospitalization | Up to 1 year
  Patients will be assessed for this outcome for up to 1 year.
Length of intensive care unit (ICU) stay | Up to 1 year
  Patients will be assessed for this outcome for up to 1 year.
Number of participants requiring mechanical ventilation | Up to 1 year
  Patients will be assessed for this outcome for up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Renumathy Dhanasekaran, MD, Principal Investigator — Stanford University
Locations (23):
- United States (23):
  - University of Arizona,, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - UCSF Fresno, Fresno, California
  - University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Georgetown University, Washington D.C., District of Columbia
  - VA Medical Center, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Medical Center, Kansas City, Kansas
  - Oschner Medical Center, Baton Rouge, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Hennepin County Medical Center (HCMC), Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kim D, Adeniji N, Latt N, Kumar S, Bloom PP, Aby ES, Perumalswami P, Roytman M, Li M, Vogel AS, Catana AM, Wegermann K, Carr RM, Aloman C, Chen VL, Rabiee A, Sadowski B, Nguyen V, Dunn W, Chavin KD, Zhou K, Lizaola-Mayo B, Moghe A, Debes J, Lee TH, Branch AD, Viveiros K, Chan W, Chascsa DM, Kwo P, Dhanasekaran R. Predictors of Outcomes of COVID-19 in Patients With Chronic Liver Disease: US Multi-center Study. Clin Gastroenterol Hepatol. 2021 Jul;19(7):1469-1479.e19. doi: 10.1016/j.cgh.2020.09.027. Epub 2020 Sep 17. PMID 32950749
- [Result] Rabiee A, Sadowski B, Adeniji N, Perumalswami PV, Nguyen V, Moghe A, Latt NL, Kumar S, Aloman C, Catana AM, Bloom PP, Chavin KD, Carr RM, Dunn W, Chen VL, Aby ES, Debes JD, Dhanasekaran R; COLD Consortium. Liver Injury in Liver Transplant Recipients With Coronavirus Disease 2019 (COVID-19): U.S. Multicenter Experience. Hepatology. 2020 Dec;72(6):1900-1911. doi: 10.1002/hep.31574. Epub 2020 Dec 9. PMID 32964510
- [Result] Adeniji N, Carr RM, Aby ES, Catana AM, Wegermann K, Dhanasekaran R. Socioeconomic Factors Contribute to the Higher Risk of COVID-19 in Racial and Ethnic Minorities With Chronic Liver Diseases. Gastroenterology. 2021 Mar;160(4):1406-1409.e3. doi: 10.1053/j.gastro.2020.11.035. Epub 2020 Nov 20. No abstract available. PMID 33227281
- [Result] Efe C, Dhanasekaran R, Lammert C, Ebik B, Higuera-de la Tijera F, Aloman C, Riza Caliskan A, Peralta M, Gerussi A, Massoumi H, Catana AM, Torgutalp M, Purnak T, Rigamonti C, Gomez Aldana AJ, Khakoo N, Kacmaz H, Nazal L, Frager S, Demir N, Irak K, Ellik ZM, Balaban Y, Atay K, Eren F, Cristoferi L, Batibay E, Urzua A, Snijders R, Kiyici M, Akyildiz M, Ekin N, Carr RM, Harputluoglu M, Hatemi I, Mendizabal M, Silva M, Idilman R, Silveira M, Drenth JPH, Assis DN, Bjornsson E, Boyer JL, Invernizzi P, Levy C, Schiano TD, Ridruejo E, Wahlin S. Outcome of COVID-19 in Patients With Autoimmune Hepatitis: An International Multicenter Study. Hepatology. 2021 Jun;73(6):2099-2109. doi: 10.1002/hep.31797. PMID 33713486